CLINICAL TRIAL: NCT03372122
Title: Evaluation of the Ability of Two Products to Remove Bacterial Spores From Subjects' Forearms
Brief Title: Removal of Bacterial Spores in Adults on Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Caroline Scott (Industry)
Responsible Party: Sponsor-Investigator, Caroline Scott, Product Claims Manager - Antiseptics, Molnlycke Health Care AB
Organization: Molnlycke Health Care AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: #170104-150
Record Dates: First submitted 2017-12-04; First posted 2017-12-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: General Skin Cleansing
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: The two study products will be assigned to opposite forearms per a computer-generated randomization schedule. Additionally, the location for baseline and post-product samples will be randomly assigned to the two longitudinally-arranged sites per forearm.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SAGE Chlorhexidine Gluconate Cloth (Active Comparator): Ready to use disinfectant cloth
  Interventions: Drug: Chlorhexidine Gluconate
- HUBS with Hibiclens (Active Comparator): Dry cloths to be used with water and disinfectant
  Interventions: Combination Product: HUBS with Hibiclens

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — A cloth to cleanse and disinfect the skin
  Arms: SAGE Chlorhexidine Gluconate Cloth
Combination Product: HUBS with Hibiclens — A dry cloth to be used in combination with water and antimicrobial soap to cleanse and disinfect the skin
  Arms: HUBS with Hibiclens

SUMMARY:
The aim of this study is to compare the effectiveness of removal of spores and dirt from the skin using a single cloth bath against a cloth bath with extra rinse step, to establish whether the extra rinse stage will lead to the removal of a higher level of spores and dirt.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the ability of two test materials to remove Clostridium difficile (ATCC #700057) spores with a tripartite soil load from subjects' forearms. For this study, removal of Clostridium difficile and the associated organic soil load will be used as an indicator of potential removal efficacy for difficult-to-remove microorganisms and associated organic matter from human skin.

All test materials are currently marketed products

ELIGIBILITY:
Inclusion Criteria:

* Subjects can be of either sex, 18 to 65 years of age, and of any race.
* Subjects must be able to read and understand English.
* Subjects must possess both forearms.
* Subjects must have healthy and short (< 1 mm in length) fingernails and cuticles with no defects. Subjects must also have no nail extensions, artificial nails, or nail polish and must not be wearing any jewelry that cannot be removed from the hands/forearms prior to testing.
* Subjects must have no tattoos, active skin rashes, dermatoses, or breaks in the skin of the hands or forearms. Subjects must also have no inflammatory skin conditions, such as atopic dermatitis / eczema or psoriasis, anywhere on the body.
* Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an organ transplant, a heart murmur, mitral valve prolapse with heart murmur, fibromyalgia, ulcerative colitis, Crohn's disease, moderate/severe asthma requiring daily use of medication, an immunocompromised condition such as AIDS (or HIV positive), lupus, or medicated multiple sclerosis.
* Subjects must read and sign the Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and List of Restricted Products prior to participating in the study.

Exclusion Criteria:

* Participation in a clinical study within 7 days of signing the informed consent for this study or current participation in another clinical study.
* Known allergies or sensitivities to latex (natural rubber), alcohols, sunscreens, deodorants, laundry detergents, inks, metals, topically-applied fragrances, cleansers, soaps, lotions, or to common antibacterial agents particularly chlorhexidine gluconate.
* Have experienced hives (raised welts) as a reaction to anything that contacted the skin.
* Use of systemic or topical antibiotic medications during either the 7-day pre-test period or on the test day.
* Use of systemic or topical steroids, other than for contraception, hormone therapy, or post-menopausal indications, during the 7-day pre-test period or on the test day. This includes steroid medications used to treat asthma.
* Have an Implanon/Nexplanon or any other dermal-implanted birth control device.
* Any prosthetic device or joint (e.g., pins, screws, plates, rods, or dental implants) anywhere in the body.
* Any type of indwelling port (or portacath) or Peripherally Inserted Central Catheter (PICC).
* Subject is pregnant, plans to become pregnant or impregnate a sexual partner within the pre-test and test periods of the study, or is nursing a child.
* Subject must not be responsible for diapering, care of wounds, intravenous management, or other bed-ridden-related care roles: have any responsibility for care of children under age 3: or be living with an immunocompromised individual.
* Any medical condition or use of any medications that, in the opinion of the Principal Investigator or consulting physician, should preclude participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Removal of Clostridium difficile and the associated organic soil load will be used as an indicator of potential removal efficacy for difficult-to-remove microorganisms and associated organic matter from human skin | 2 hours
  As a measure of the ability of the test materials to remove spores from the skin, reductions will be calculated by subtracting the population of spores recovered from a treated sites from the population recovered from the baseline sites.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Griggs, M.S, CCRC, Principal Investigator — BSLI
Locations (1):
- Bioscience Laboratories, Inc, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided